CLINICAL TRIAL: NCT02002455
Title: Preoperative Staging and Dose Escalated Radiotherapy of Prostate Carcinoma
Brief Title: Preoperative Staging and Dose Escalated Radiotherapy of Prostate Carcinoma With PET and MRI
Acronym: Flucipro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: GE Healthcare (Industry); Blue Earth Diagnostics (Industry)
Responsible Party: Principal Investigator, Heikki Minn, Professor, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T70/2013
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Carcinoma
Keywords: FACBC; PET/CT; PET/MRI; Radical prostatectomy; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography; Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multimodality imaging (Experimental): PET/CT, PET/MRI, mpMRI
  Interventions: Device: PET/CT, PET/MRI, mpMRI

INTERVENTIONS:
Device: PET/CT, PET/MRI, mpMRI — FACBC dose 370 megabecquerel (MBq)

SUMMARY:
Prostate cancer (PCa) is currently the most common neoplastic disease among men in well-developed countries with 350 000 new cases diagnosed annually in Europe and 4 800 in Finland. Due to widespread use of serum prostate specific antigen (PSA) in asymptomatic men, most patients present initially with localized disease. Radical prostatectomy, radiotherapy (RT) and active surveillance are the most common management options for patients with localized PCa. Proper preoperative staging for patients with adverse features on biopsy who are candidates for radical prostatectomy is urgently needed. For elderly men external beam RT is the preferred modality which can be safely performed utilizing modern techniques such as intensity modulated and image guided radiotherapy (IMRT and IGRT). Since randomized studies suggest a dose response effect beyond 78-80 Gy newer techniques aim at dose escalation provided that toxicity can be controlled. Therefore, ultra high dose IMRT/IGRT requires visualization of intracapsular disease which will receive the highest dose. Taken together, the use of accurate anatomical and functional imaging modalities are essential for planning both nerve sparing radical prostatectomy and ultra high dose IMRT/IGRT Fluorine-18 labeled L-leucine analogue 1-amino-3-fluorocyclobutane-1-carboxylic acid (FACBC) has shown to preferentially accumulate in PCa and its nodal metastases. By assisting in localization of intraprostatic and pelvic disease FACBC with hybrid positron emission tomography/computed tomography (PET/CT) or magnetic resonance imaging (PET/MRI) has potential to improve selection of patients for robot-assisted radical prostatectomy and IMRT/IGRT.

Anatomical MRI at 1.5 Tesla (T) compared with transrectal ultrasound has demonstrated a higher sensitivity for tumor detection but almost the same specificity, stressing the need for additional metabolic MRI. Advanced application of MRI such as proton magnetic resonance spectroscopy (1H MRS), diffusion weighted imaging (DWI) and dynamic contrast enhanced imaging (DCE-MRI) are increasingly being used for detection and characterization of PCa. The use of 3T scanners and multiparametric MRI (mpMRI), consisting of anatomical MRI, DWI, 1H MRS and DCE-MRI, demonstrated very promising result for staging and detection of PCa.

DETAILED DESCRIPTION:
Specific aims of the current study are as follows:

i) To determine the sensitivity, specificity and accuracy of multiparametric 3T MRI, (anatomical MRI, DCE-MRI, DWI and 1H MRS) combined with FACBC PET/CT and PET/MRI in correlation with systematic biopsy and whole mount prostatectomy specimens.

ii) To asses the applicability of multiparametric 3T MRI combined with FACBC-PET/CT and PET/MRI for detection of cancer aggressiveness based on Gleason score and PSA.

iii) To develop quantitative and qualitative methods for evaluation of FACBC PET/MRI

iv) To develop and validate an imaging protocol which will become the standard protocol for prostate imaging both for surgical and radiotherapy patients at Turku PET Centre using hybrid PET/MRI

ELIGIBILITY:
Inclusion Criteria:

* Age: 50 to 85 years old
* Language spoken: Finnish or Swedish
* Diagnosis: Histologically confirmed adenocarcinoma of prostate
* Adequate histological sampling consisting of at least 3 biopsy samples from each lobe
* No previous surgical, radiation or endocrine treatment for prostate carcinoma
* Clinical stage T1c-T3aN0 based on transrectal ultrasound
* Serum creatinine ≤ 1,5 x upper limit of normal (ULN)
* Patient agrees to undergo either surgery or external radiotherapy
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Prior medical history: Patient must have no history of serious cardiovascular, liver or kidney disease
* Infections: Patient must not have an uncontrolled serious infection
* No contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* Patient preference for active surveillance as a method of prostate cancer management

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of hybrid PET/MRI with FACBC | 1 years
  By comparing tracer uptake and imaging findings at MRI in each sextant with macroslices obtained at radical prostatectomy sensitivity, specificity, positive and negative predictive value and accuracy will be calculated

SECONDARY OUTCOMES:
Biochemical relapse free survival (bRFS) | 5 years
  By sequential measurements of serum PSA bRFS will be determined in patients having biologically guided radiotherapy (BGRT) plans. BGRT is performed with dose painting of hot spots at PET/MRI

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Minn, Professor, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jambor I, Kuisma A, Kahkonen E, Kemppainen J, Merisaari H, Eskola O, Teuho J, Perez IM, Pesola M, Aronen HJ, Bostrom PJ, Taimen P, Minn H. Prospective evaluation of 18F-FACBC PET/CT and PET/MRI versus multiparametric MRI in intermediate- to high-risk prostate cancer patients (FLUCIPRO trial). Eur J Nucl Med Mol Imaging. 2018 Mar;45(3):355-364. doi: 10.1007/s00259-017-3875-1. Epub 2017 Nov 16. PMID 29147764